CLINICAL TRIAL: NCT04951557
Title: Setting Benchmarks for Transsphenoidal Resection of Pituitary Adenomas - An Analysis of Standardized Outcome References From an International Multicentre Cohort
Brief Title: Setting Benchmarks for Transsphenoidal Resection of Pituitary Adenomas
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Richard Drexler, Principal Investigator, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: Benchpit
Record Dates: First submitted 2021-06-17; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-06

CONDITIONS: Pituitary Adenoma; Pituitary Tumor; Pituitary Diseases
MeSH Terms: conditions — Pituitary Neoplasms; Pituitary Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Transsphenoidal resection — Transsphenoidal resection of pituitary adenoma

SUMMARY:
To conduct a retrospective multicenter cohort study to define benchmark values for best achievable outcomes following transsphenoidal resection of pituitary adenomas.

DETAILED DESCRIPTION:
Surgeons strive for the best possible outcome of their surgeries with the greatest possible chance for recovery of the patients. Therefore, monitoring and quality improvement is increasingly important in surgery. For this purpose, different concepts were developed with the aim to assess best achievable results for several surgical procedures and reduce unwarranted variation between different centers. The concept of a benchmark establishes reference values which represents the best possible outcome of high-volume centers and can be used for comparison and improvement. In the past years, the concept of benchmarking attaches greater importance in the field of healthcare, especially in surgery. Benchmark values are established within a patients' cohort for which the best possible outcome can be expected. To date, no valid concept exists to describe the outcome of patients after transsphenoidal resection of pituitary adenomas. The aim of our study is the establishment of robust and standardized outcome references after transsphenoidal surgery. After successful implantation of benchmarks from an international cohort of renowned centers, these data serve as reference values for the evaluation of novel surgical techniques and comparisons among centers or future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients who went through transsphenoidal resection of pituitary adenoma
* Including high-volume centres with ≥50 cases per year

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who went through transsphenoidal resection of pituitary adenoma at high-volume centres
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2017-01-31 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Reoperation | up to two weeks
CSF leak | up to two weeks
  Requiring intervention
Epistaxis | up to two weeks
  Requiring intervention
Meningitis | up to two weeks
Diabetes insipidus | up to two weeks
SIADH | up to two weeks
Cerebral vasospasm | up to two weeks
New hypopituitarism | up to two weeks
  Requiring hormone replacement
Normalization of hormone levels | up to two weeks
New neurological deficit | up to two weeks
Postoperative change of vision | up to two weeks
Need for ICU care | up to two weeks
Length of stay | up to two weeks
In-hospital mortality | up to two weeks
Readmission to hospital | At 6 months follow up
  Related to transsphenoidal surgery
Electrolyte imbalance | At 6 months follow up
  Requiring drug treatment
New hypopituitarism | At 6 months follow up
  Requiring hormone replacement
New neurological deficit | At 6 months follow up
CSF leak | At 6 months follow up
  Requiring intervention
Termination of hypersecretion | At 6 months follow up
  If applicable
MRI resection control | At 6 months follow up
  If applicable

OTHER OUTCOMES:
Age | At time of surgery
Gender | At time of surgery
Body mass index | At time of surgery
ASA score | At time of surgery
Hormone replacement | At time of surgery
Neurological deficit | At time of surgery
Previous therapy | At time of surgery
  None, transsphenoidal surgery, pharmacotherapy, radiotherapy
Tumour size | At time of surgery
  Microadenoma, Macroadenoma
Knosp grade | At time of surgery
Tumour extension | At time of surgery
  Intraventricular extension, sinus cavernous invasion
Histology | At time of surgery
  According to 2017 WHO classification
Operating method | Surgery
  Endoscopy, microscopy, 3D-video microscopy, hybrid
Operating duration | Surgery
  minutes
Gross total resection | Surgery
Blood transfusion | Surgery
Repair of CSF leak | Surgery
  None, muscle/fascial patch, fibrin alone, mucosal flap, fat, other technique
Nasal tamponade | Surgery

CONTACTS AND LOCATIONS:
Overall Officials: Richard Drexler, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf; Franz L Ricklefs, MD, Principal Investigator — Universitätsklinikum Hamburg-Eppendorf; Jörg Flitsch, MD, Study Chair — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Undecided